CLINICAL TRIAL: NCT00998972
Title: Preventive Administration of N-acetyl-cysteine (NAC) in Organ Donor: Effects on Kidney Graft Function
Brief Title: N-acetyl-cysteine (NAC) and Kidney Graft Function
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institut d'Anesthesiologie des Alpes Maritimes (Other)
Responsible Party: Carole Ichai, Institut d'Anesthésiologie des AM
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NAC-CHUN1
Record Dates: First submitted 2009-10-17; First posted 2009-10-21 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2009-06

CONDITIONS: Brain Death; Chronic Renal Insufficiency
Keywords: kidney graft,; delayed graft function; N-acetylcysteine
MeSH Terms: conditions — Brain Death; Renal Insufficiency, Chronic; Delayed Graft Function | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- control (No Intervention): control arm without any specific intervention
- N-acetylcysteine (Experimental): administration of 600 mg intravenous N-acetyl cysteine before and 2 hours after angiography performed for the diagnosis of brain death
  Interventions: Drug: N-acetylcysteine

INTERVENTIONS:
Drug: N-acetylcysteine — 600 mg intravenous before and 2 hours after cerebral arteriography
  Other Names: n-acetylcysteine administration
  Arms: N-acetylcysteine

SUMMARY:
The goal of this study is to evaluate the effect of N-acetyl-cysteine (NAC) administration in organ donors on the kidney graft function of recipients.

DETAILED DESCRIPTION:
Ischemia-reperfusion is a major contributing factor for delayed renal function after transplantation. It has been shown that the administration of an antioxidant, i.e. NAC, in patients with chronic renal insufficiency may prevent radio contrast-induced nephropathy. Due to its antioxidant effects, organ donor pretreatment with NAC has demonstrated to improve renal graft function in two experimental studies. Study objectives: to compare the incidence of delayed graft renal function between two groups of patients, i.e., those receiving the graft from organ donors pretreated with NAC and a group control. The primary endpoint was the number of delayed graft function defined as the requirement of at least one sequence of dialysis during the first seven days following transplantation. Secondary endpoints: evolution of creatininemia, azotemia at day 1, 7, 14 and ,30 after surgery; acute and delayed transplant rejection; intrahospital mortality.

Patients inclusion: all organ donors and recipients were eligible Exclusion criteria: for organ donors were preexistent chronic renal insufficiency and contra-indications for kidney procurement; for recipient were transplantation outside our hospital The donors were randomized in a single-blind fashion into two groups : the control group and the group receiving 600 mg IV of NAC 1 hour before and 600 mg IV 2 hours after cerebral arteriography required to diagnose brain death. Sample size has been calculated delayed graft function by 50% leading to include 118 recipients in each group.

Follow up: one year after transplantation. Study beginning in september 2006. Length of inclusion during 36 months.

ELIGIBILITY:
Inclusion Criteria:

* all recipient for kidney graft in our hospital

Exclusion Criteria:

* transplantation out side our hospital
* refusal from the patient

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2006-09; Primary Completion 2010-12 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Incidence of delayed graft function | 1 year

SECONDARY OUTCOMES:
Evolution of creatininemia and azotemia during the first month after transplantation | 30 days
Intrahospital mortality | 30 days
Acute and delayed graft rejection | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Carole R Ichai, MD, PhD, Principal Investigator — Service de Reanimation Medicochirurgical. CHU de Nice
Locations (1):
- CHU de Nice, Nice, Alpes Maritimes, France

REFERENCES:
- [Derived] Colombijn JM, Hooft L, Jun M, Webster AC, Bots ML, Verhaar MC, Vernooij RW. Antioxidants for adults with chronic kidney disease. Cochrane Database Syst Rev. 2023 Nov 2;11(11):CD008176. doi: 10.1002/14651858.CD008176.pub3. PMID 37916745
- [Derived] Orban JC, Quintard H, Cassuto E, Jambou P, Samat-Long C, Ichai C. Effect of N-acetylcysteine pretreatment of deceased organ donors on renal allograft function: a randomized controlled trial. Transplantation. 2015 Apr;99(4):746-53. doi: 10.1097/TP.0000000000000395. PMID 25250647